CLINICAL TRIAL: NCT04833114
Title: Open-label, Prospective Phase III Clinical Study to Compare Polatuzumab Vedotin Plus Rituximab, Ifosfamide, Carboplatin and Etoposide (Pola-R-ICE) With Rituximab, Ifosfamide, Carboplatin and Etoposide (R-ICE) Alone as Salvage Therapy in Patients With Primary Refractory or Relapsed Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Polatuzumab Vedotin Plus Rituximab, Ifosfamide, Carboplatin and Etoposide (Pola-R-ICE) Versus R-ICE Alone in Second Line Treatment of Diffuse Large B-cell Lymphoma (DLBCL)
Acronym: Pola-R-ICE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pola-R-ICE; MO40599 / GLA 2017-R2 (Other: Financier)
Record Dates: First submitted 2021-02-10; First posted 2021-04-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Diffuse Large B-cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Rituximab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm: Pola-R-ICE (Experimental): combination of standard chemotherapy with polatuzumab vedotin (Pola-R-ICE) Application
  Interventions: Drug: Polatuzumab Vedotin; Drug: Mabthera; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide
- Standard Arm: R-ICE (Active Comparator): conventional treatment with rituximab, ifosfamide, carboplatin and etoposide (R-ICE)
  Interventions: Drug: Mabthera; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Polatuzumab vedotin 1.8 mg/kg will be administered intravenously on Day 1 of each 21-day cycle for up to 3 cycles.
  Arms: Experimental Arm: Pola-R-ICE
Drug: Mabthera — Rituximab (Mabthera/Rituxan®) will be administered as per local practice at a dose of 375 mg/m2 intravenously on Day 1 of each 21-day cycle for up to 3 cycles.
Drug: Ifosfamide — Ifosfamide 5000 mg/m² will be administered i.v. over a 24 hr period starting on cycle Day 2.
Drug: Carboplatin — Carboplatin AUC 5 max 800 mg will be administered i.v. on cycle Day 2.
Drug: Etoposide — Etoposide 100 mg/m² will be administered i.v. on cycle Days 1, 2 and 3.

SUMMARY:
An open-label, prospective Phase III clinical study to compare polatuzumab vedotin plus rituximab, ifosfamide, carboplatin and etoposide (Pola-R-ICE) with rituximab, ifosfamide, carboplatin and etoposide (R-ICE) alone as salvage therapy in patients with primary refractory or relapsed diffuse large B-cell lymphoma (DLBCL)

DETAILED DESCRIPTION:
The study is designed as an international, multicenter, open-label, two-arm, prospective phase III study to compare the treatment of polatuzumab vedotin plus rituximab, ifosfamide, carboplatin and etoposide (Pola-R-ICE) with the combination of rituximab, ifosfamide, carboplatin and etoposide (R-ICE) alone as salvage therapy in patients with primary refractory or relapsed DLBCL.

The study will involve study sites in Germany, UK, Spain, and Austria. It is planned to include 324 patients who will be randomized 1:1 to receive either treatment in the experimental arm (Pola-R-ICE) or in the standard arm (R-ICE) to end up with 308 evaluable subjects for the randomized part of the trial. Further 10 patients will be treated with Pola-R-ICE during the safety run-in phase.

The study consists of a screening/inclusion visit, three chemotherapy cycles, an end-of - treatment visit (EoT), and follow-up visits. For each subject, the total duration of the study will be approximately 3 months of treatment plus at least 21 months follow-up. The study will end when the last included patient will have passed the last follow-up visit (LPLFU). For the study as a whole, the primary outcome will be evaluated when the last included patient will have completed the 21 months follow-up period or has left the study prematurely.

For the study as a whole, the primary outcome will be evaluated when the last included patient will have completed the 21 months follow-up period or has left the study prematurely.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent form must be signed before any study specific tests or procedures are done
2. Adult male and female patients ≥18 years (≥16 years in the UK*) at the time of inclusion in the study (* In the UK an "adult" means a person who has attained the age of 16 years, according to The Medicines for Human Use (Clinical Trials) Regulations 2004, Part 1 Point 2.)
3. Ability to understand and follow study-related instructions
4. Risk group: All patients with one of the following histologically defined entities: Histological diagnosis of primary refractory or relapsed aggressive B-cell non-Hodgkin lymphoma (B-NHL), confirmed by a biopsy of involved nodal or extranodal site. Patients with any of the following histologies can be included:

   * DLBCL not otherwise specified (NOS)
   * T-cell/histiocyte-rich large B-cell lymphoma
   * Primary cutaneous DLBCL, leg type
   * Epstein-Barr virus (EBV)-positive DLBCL, NOS
   * DLBCL associated with chronic inflammation
   * Primary mediastinal (thymic) large B-cell lymphoma
   * High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements
   * High-grade B-cell lymphoma, NOS

   Refractory disease is defined as no complete remission to first line therapy; subjects who are intolerant to first line therapy are excluded. Three groups of patients are eligible:
   * Progressive disease (PD) as best response to first line therapy (biopsy not mandatory if diagnostic sample available).
   * Stable disease (SD) as best response after at least 4 cycles of first line therapy (e.g., 4 cycles of R-CHOP) (biopsy not mandatory if diagnostic sample available).
   * Partial response (PR) as best response after at least 6 cycles, and biopsy-proven residual disease or disease Progression after the partial response.

   Relapsed disease is defined as complete remission to first line therapy followed by biopsy proven disease relapse.
5. Performance Status ECOG 0-2 at time of randomization or ECOG 3 at screening if this is DLBCL-related and has improved to ECOG 2 or less with a 7-day steroid treatment during the screening Phase (e.g. 1 mg/kg prednisone).
6. Information on all 5 International Prognostic Index (IPI) factors
7. Staging (PET-CT based-staging according to Lugano criteria 2014). Patients must have PET-positive lesions.
8. Subjects must have received adequate first line therapy including at a minimum: i) anti-CD20 monoclonal antibody unless Investigator determines that tumor is CD20 negative, and ii) an anthracycline containing chemotherapy Regimen
9. Intent to proceed to high-dose therapy (HDT) and stem cell transplantation (SCT) if response to second line therapy
10. Adequate hematological function, as defined by: hemoglobin ≥ 8 g/dL, absolute neutrophil count (ANC) ≥ 1.0 x 109/L OR ≥ 0.5 x 109/L if neutropenia is attributable to underlying disease and before the administration of steroids, and platelet count ≥ 75 x 109/L OR ≥ 50 x 109/L if thrombocytopenia is attributable to Underlying disease
11. Women of childbearing potential must have a negative pregnancy test result within 7 days prior to the first study drug Administration
12. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs
13. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

(1) Serious accompanying disorder leading to impaired organ function causing significant clinical problems and reduced life expectancy of less than 3 months. In particular, patients with the following organ dysfunction caused by accompanying disorders are to be excluded:

* Heart failure with left ventricular ejection fraction (LVEF) < 45%
* Impaired pulmonary function with vital capacity (VC) or forced expiratory volume (FEV1) < 50% of normal (only in case of history of significant pulmonary disease)
* Impaired renal function with glomerular filtration rate (GFR) < 50 mL/min (calculated)
* Impaired liver function with alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT) or Bilirubin > 1.5 x upper limit of normal (ULN). If elevation is caused by the disease, threshold of 2.5 x ULN is accepted
* Peripheral neuropathy > Grade II (2) Human immunodeficiency virus (HIV)-positivity with detectable viral load and/or a CD4+ count below 0.3/nL

  (3) Hepatitis B and C as defined by seropositivity (HBsAG and anti HBe/ anti HBc; anti-Hc); in case of false positive serology (transfused antibodies) negative PCR-results will allow patient inclusion. Patients with occult or prior HBV infection (defined as negative HBsAg and positive hepatitis B core antibody [HBcAb]) may be included if HBV DNA is undetectable, provided that they are willing to undergo DNA testing on Day 1 of every cycle and monthly for at least 12 months after the last cycle of study Treatment

  (4) Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study inclusion or any unresolved major episode of infection (as evaluated by the investigator) within 1 week prior to Cycle 1 Day 1

  (5) Patients with suspected or latent tuberculosis. Latent tuberculosis needs to be confirmed by positive interferon-gamma release Assay

  (6) Primary or secondary central nervous system (CNS) lymphoma at the time of recruitment

  (7) Richter's transformation or prior chronic lymphocytic leukemia (CLL)

  (8) Vaccination with a live vaccine within 4 weeks prior to Treatment

  (9) Recent major surgery (within 6 weeks before the start of Cycle 1 Day 1) other than for diagnosis

  (10) Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to Cycle 1 Day 1

  (11) Received more than one line of therapy for DLBCL

  (12) Received polatuzumab vedotin as part of the first line therapy

  (13) Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

  (14) Ongoing treatment or study procedures within any other Investigational Medicinal Product (IMP) clinical trial with the exception of follow-up. In case of a preceding clinical trial, last application of the respective IMP(s) must have been done more than five elimination half-lives before start of study medication in this trial.

  (15) History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies

  (16) History of hypersensitivity to any of the study drugs or their ingredients or to drugs with similar structure

  (17) Contraindications according to the Investigator´s Brochure (IB) of polatuzumab vedotin or the local Summary of Product Characteristics (SmPCs) of the used rituximab, ifosfamide, carboplatin or etoposide products

  (18) Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's Safety

  (19) Pregnancy or breastfeeding, or intending to become pregnant during the study or within 12 months after the last dose of study drug

  (20) Close affiliation with the investigator (e.g. a close relative) or persons working at the study site

  (21) Subject is an employee of the sponsor or involved Contract Research Organization

At study inclusion, any organ impairment due to lymphoma infiltration is NOT regarded as an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the event-free survival of patients with DLBCL at first progression and the occurrence of any of the following events: | Day of randomization until end of follow up (12 weeks treatment and at least 21 months follow up)
  * Failure to achieve sufficient response in PET-CT (Deauville score 3 or less) at end of study treatment (metabolic CR)
  * Disease progression (PD)
  * Start of additional unplanned anti-tumor treatment (radiation therapy allowed)
  * Relapse after achieving CR
  * Death due to any cause

SECONDARY OUTCOMES:
Assessment of the rate of metabolic complete response. | Day of randomization until end weeks 12 treatment.
  Number of complete remissions.
Evaluation of the partial response rate. | Day of randomization until end of 12 weeks treatment.
  Number of partial responses.
Assessment of the overall response rate. | Day of randomization until end of 12 weeks treatment.
  Number of complete and partial responses.
Assessment duration of response. | Day of randomization until end of follow up (12 weeks treatment and at least 21 months follow up)
  Time from documentation of tumor response to disease progression or relapse.
Assessment of the rate of progressive disease. | Day of randomization until end of 12 weeks treatment.
  Number of progressive diseases.
Assessment of disease relapse. | Day of randomization until end of 12 weeks treatment.
  Number of relapses.
Assessment of progression free survival. | Day of randomization until end of follow up (12 weeks treatment and at least 21 months follow up)
  Occurence of disease progression, relapse or death due to any cause.
Assessment of overall survival. | Day of randomization until end of follow up (12 weeks treatment and at least 21 months follow up)
Assessment of the rate of patients proceeding to transplantation. | Day of randomization until week 12.
Assessment of the rate of patients with non-relapse mortality. | Day of randomization until end of follow up (12 weeks treatment and at least 21 months follow up)
Evaluation of the frequency of adverse and serious adverse events including the incidence and duration of the adverse events neutropenia and thrombocytopenia with grade 4. | Day of Randomization until 28 days after start of last cycle or start of further therapy
Assessment of the number of patients with treatment-related death. | Day of Randomization until up week 12 or 2 months after week 12 but before start of further therapy
To determine the number of patients with occurence of second malignancies | Day of Randomization until Day of randomization until end of follow up (at least 21 months follow up)
Assessment of the protocol adherence by the rate and duration of chemotherapy cycles patients received. | Day of Randomizaton until week 12.
Assessment of the cumulative and relative dose of each IMP( ifosfamide, carboplatin and etoposide, rituximab and of the polatuzumab vedotin) by quantitative measurement. | Day of Randomizaton until week 12.
Assessment of the change in health related quality of life by generic questionnaire. | Day of Randomization until weeks 12 and months 3 and 12 in follow up.
  Scale scores to be obtained for the multi-items scales. Range in score from 0 to 100. A high scale score represents a higher response level.
Assessment of the change in health related quality of life by five-item questionnaire. | Day of Randomization until weeks 12 and months 3 and 12 in follow up
Assessment visual analogue scale to measure health state. | Day of Randomization until weeks 12 and months 3 and 12 in follow up
  This scale is provided with numbers from 0 to 100.100 is the best health state and 0 (zero) is the worst health state.
Functional assessment of the cancer therapy-lymphoma by general questions and specific questions for lymphoma. | Day of Randomization until weeks 12 and months 3 and 12 in follow up.
  Assessment how lymphoma-specific symptoms impact quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Glaß, Prof., Principal Investigator — HELIOS Klinik Berlin-Buch, Klinik für Hämatologie und Stammzelltransplantation
Locations (64):
- Austria (8):
  - UK Graz Universitätsklinik für Innere Medizin Klinische Abteilung für Hämatologie, Graz
  - LKH Hochsteiermark Standort Leoben Abteilung für Innere Medizin Department für Hämato-Onkologie, Leoben
  - Ordensklinikum Linz GmbH- Elisabethinen: I. Interne Abteilung Hämato-Onkologie, Linz
  - Kepler Universitätsklinikum Med Campus III, Univ.-Klinik für Hämatologie und Internistische Onkologie, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - AKH Meduni Wien Universitätsklinik für Innere Medizin I:, Vienna
  - Hanusch Krankenhaus, Vienna
  - Klinikum Wels-Grieskirchen Abteilung für Innere Medizin IV, Wels
- Germany (26):
  - Universitätsklinikum RWTH-Aachen, Aachen
  - HELIOS Klinik Berlin-Buch, Klinik für Hämatologie und Stammzelltransplantation, Berlin
  - Städtisches Klinikum Braunschweig, Braunschweig
  - DIAKO Ev.Diakonie-Krankenhaus gemeinnützige GmbH, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - St. Johannes Hospital Dortmund, Dortmund
  - Universitätsklinikum Dresden, Dresden
  - Helios St. Johannes Klinik, Duisburg
  - Klinik für Onkologie, Hämatologie und Palliativmedizin, Düsseldorf
  - Universitätsklinikum Frankfurt, Frankfurt
  - Georg-August-Universität Göttingen Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Städtisches Krankenhaus Kiel, Kiel
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Philipps-Universität Marburg, Marburg
  - Universitätsklinikum Münster, Münster
  - Klinikum Oldenburg, Oldenburg
  - Unversitätsmedizin Rostock, Rostock
  - Klinikum Stuttgart, Stuttgart
  - Klinikum Mutterhaus, Trier
  - Universitätsklinikum Ulm, Ulm
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Spain (21):
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Universitario de Cabueñes, Gijón
  - Institut Català d'oncologia de L'Hospitalet (ICO-L'Hospitalet), L'Hospitalet de Llobregat
  - Complejo Hospitalario Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Clínica Universidad de Navarra (Madrid location), Madrid
  - Hospital Universitario Fundación Jimenez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Clínica Universidad de Navarra (Pamplona location), Pamplona
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
- United Kingdom (9):
  - Belfast City Hospital, Belfast
  - Royal Cornwall Hospital, Cornwell
  - St James University Hospital, Leeds
  - University London College Hospitals, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth, Plymouth
  - Queens Hospital, Romford, Romford
  - University Hospital Southampton NHS, Southampton